CLINICAL TRIAL: NCT01725607
Title: Postoperative Sleep Quality in Patients Undergoing Thoracic Surgery With Different Types of Anesthesia Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, associate professor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20121101
Record Dates: First submitted 2012-11-03; First posted 2012-11-14 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2013-10

CONDITIONS: General Anesthesia, Thoracic Epidural Anesthesia
Keywords: dexmedetomidine, thoracic epidural anesthesia
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- the control group (Group C) (No Intervention): general anesthesia
- general anesthesia combined with dexmedetomidine infusion (Experimental): general anesthesia combined with 1 μg/kg dexmedetomidine infusion after induction (Group D)
  Interventions: Drug: general anesthesia combined with dexmedetomidine infusion
- general anesthesia combined with TEA (Experimental): general anesthesia combined with TEA (Group E)
  Interventions: Procedure: general anesthesia combined with TEA

INTERVENTIONS:
Drug: general anesthesia combined with dexmedetomidine infusion — general anesthesia combined with 1 μg/kg dexmedetomidine infusion after induction (Group D)
  Arms: general anesthesia combined with dexmedetomidine infusion
Procedure: general anesthesia combined with TEA — general anesthesia combined with TEA (Group E)
  Arms: general anesthesia combined with TEA

SUMMARY:
We designed a study to determine whether a single dose of dexmedetomidine or thoracic epidural anesthesia combined with general anesthesia would provide hemodynamic stability, reduce stress hormone responses, inhibit inflammatory cytokine secretion, and improve sleep quality in patients after thoracic surgery.

DETAILED DESCRIPTION:
We designed a prospective, single-blinded, randomized, and controlled study to determine whether a single dose of dexmedetomidine or thoracic epidural anesthesia combined with general anesthesia would provide hemodynamic stability, reduce stress hormone responses, inhibit inflammatory cytokine secretion, and improve sleep quality in patients after thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* lung surgery
* one-lung ventilation.

Exclusion Criteria:

* body mass index exceeding 30 kg/m2,
* autonomic dysfunction,
* cardiovascular disease,
* neurological or psychiatric diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
inflammatory cytokine secretion and postoperative sleep quality | immediately before anesthesia (T1), 5 min after endotracheal intubation (T2), immediately after incision (T3), 5 min after OLV initiation (T4), 5 min after double-lung ventilation initiation (T5), and immediately after extubation (T6)
  Primary outcomes were inflammatory cytokine secretion and postoperative sleep quality, which was measured with the BIS data on first and second postoperative nights.

SECONDARY OUTCOMES:
amine secretion during the surgical period and hemodynamic stability | immediately before anesthesia (T1), 5 min after endotracheal intubation (T2), immediately after incision (T3), 5 min after OLV initiation (T4), 5 min after double-lung ventilation initiation (T5), and immediately after extubation (T6)
  amine (epinephrine and norepinephrine) secretion during the surgical period and hemodynamic stability

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ma, M.D.,PhD., Study Chair — Dept. of Anesthesiology, the First Hospital of CMU
Locations (1):
- Department of Anesthesiology, the First Hospital of China Medical University, Shenyang, Liaoning, China